CLINICAL TRIAL: NCT00715364
Title: A Phase IIb Prospective, Randomized, Double-blind, Placebo Controlled Study of NTx™-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients
Brief Title: REGENESIS (US): A Phase IIb Prospective, Randomized, Double-blind, Placebo Controlled Study of NTx™-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients
Acronym: REGENESIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Stem Cell Therapeutics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTx™-265-CP-201-IS (US)
Record Dates: First submitted 2008-07-09; First posted 2008-07-15 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Ovidrel; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: NTx™-265: rhCG, then rEPO
- 2 (Placebo Comparator)
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: NTx™-265: rhCG, then rEPO — * rhCG 385 µg, SC, on Day 1, 3, and 5 of study participation, then
  * rEPO 30,000 IU, IV, on Day 7, 8, and 9 of study participation
  Other Names: Ovidrel; Epogen
  Arms: 1
Drug: Saline Placebo — * Saline SC, on Day 1, 3, and 5 of study participation, then
  * Saline IV, on Day 7, 8, and 9 of study participation
  Other Names: Sodium Chloride 0.9%
  Arms: 2

SUMMARY:
To assess the safety and tolerability of NTx™-265 when given to acute ischemic stroke patients.

To assess the neurological outcome in acute ischemic stroke patients treated with NTx™-265, when compared with patients given a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85.
* NIHSS score 6-24 within 24-48 hours after stroke onset and enrolment.
* Stroke is ischemic in origin, supratentorial, and radiologically confirmed (CT scan or diagnostic MRI) prior to enrolment.
* Patient is 24-48 hours from time of stroke onset when the first dose of NTx™-265 therapy is administered. Time of onset is when symptoms began; for stroke that occurred during sleep, time of onset is when patient was last seen or was self-reported to be normal.
* Reasonable expectation of availability to receive the full 9 day NTx™-265 course of therapy, and to be available for subsequent follow-up visits.
* Reasonable expectation that patient will receive standard post-stroke physical, occupational, speech, and cognitive therapy as indicated.
* Female patient is either:

  1. not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or,
  2. if of childbearing potential, agrees to use two of the following effective separate forms of contraception throughout the study, up to and including the follow up visits: i) condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD) contraceptives (e.g. implants, injectables, combined oral, etc.) OR ii) a vasectomized partner OR iii) abstinence

Exclusion Criteria:

* Patients presenting with lacunar, hemorrhagic and/or brain stem stroke
* Patients classified as comatose, defined as a patient who requires repeated stimulation to attend, or is obtunded and requires strong or painful stimulation to make movements (NIHSS 1A score must be <2)
* Women who have tested positive for pregnancy, or are breast-feeding, or are not using a highly effective method of birth control that can be maintained for the duration of the study
* Serum hemoglobin > 16 g/dL (males) or > 14 g/dL (females); or platelet count > 400,000/mm3
* Advanced liver, kidney, cardiac, or pulmonary disease; the former will be operationally defined using NCI Toxicity Criteria (Grade 2 or higher)
* Serum bilirubin > 1.5 x ULN
* Alkaline phosphatase > 2.5 x ULN
* AST or ALT > 2.5 x ULN
* Creatinine > 2.0 x ULN
* Patients with known and documented Transferrin saturation <20% or ferritin < 100 ng/ml
* Patients with known and documented elevated PSA levels
* Patients with a known history of hypercoagulability, including known cardiolipin/antiphospholipid antibody syndrome
* Expected survival < 1 year
* Allergy or other contraindication to hCG
* Allergy or other contraindication to epoetin alfa:
* A known diagnosis of cancer (except non-malignant skin cancer)
* Uncontrolled hypertension, defined in the context of acute stroke as blood pressure persistently above 220 mm Hg systolic or 120 mm Hg diastolic despite antihypertensive therapy
* Use of either hCG or epoetin alfa within the previous 90 days
* Any condition known to elevate hCG, active in the prior 24 months, e.g., choriocarcinoma or germ cell tumor
* Patients with a pre-stroke/pre-morbid modified Rankin Score (mRS) ≥ 2
* Any patients living in a nursing home or supervised living center. Patients must be historically fully independent in all activities of daily living including banking, shopping, cooking, toileting, showering and dressing
* Any other medical condition or degree of stroke such that, in the investigator's opinion, the patient should not be included in the trial
* With the exception of the qualifying stroke, any other stroke within the previous 3 months
* Patients who cannot take anti-platelet or anti-coagulant therapy
* Pre-existing and active major psychiatric or other chronic neurological disease
* Consume, on average, greater than 14 alcoholic drinks per week, or have a history of substance abuse or dependency within 12 months prior to the study
* Currently participating in another investigational study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events | screening to Day 90

SECONDARY OUTCOMES:
mRS | Day 90
NIHSS | Day 90
Barthel Index | Day 90
Action Research Arm Test | Day 90
Gait Velocity Test | Day 90
Boston Naming Test | Day 90
Line Cancellation Test | Day 90
Trails A & B Test | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Cramer, MD, MMSc, Principal Investigator — Department of Neurology, University of Califonia, Irvine Medical Center
Locations (2):
- United States (2):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California, Irvine Medical Center, Orange, California